CLINICAL TRIAL: NCT01348386
Title: Efficacy and Tolerance of the Topical Application of Potassium Hydroxide (10% and 15%) in the Treatment of Molluscum Contagiosum
Brief Title: Efficacy and Tolerance of Potassium Hydroxide (10% and 15%) in Molluscum Contagiosum
Acronym: EKOH-MOL 2008
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC08/00011
Record Dates: First submitted 2011-05-04; First posted 2011-05-05 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2011-05

CONDITIONS: Molluscum Contagiosum
Keywords: Potassium hydroxide.; Molluscum Contagiosum
MeSH Terms: conditions — Molluscum Contagiosum | interventions — potassium hydroxide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- KOH 10% (Experimental): Treatment consists of the application of topical 10% KOH in an aqueous solution.
  Interventions: Drug: Hydroxide Potassium
- KOH 15% (Experimental): Treatment consists of the application of topical 15% KOH in an aqueous solution
  Interventions: Drug: Hydroxide Potassium
- PLACEBO (Placebo Comparator): 100 milliliters of saline solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxide Potassium — Treatment will consist of the application of topical 10% or 15% KOH in an aqueous solution for the two treatment groups, compared to a placebo-treated control group. Topical Application.
  Arms: KOH 10%; KOH 15%
Drug: Placebo
  Arms: PLACEBO

SUMMARY:
BACKGROUND:

Molluscum contagiosum is a non-serious children viral infection. Because of its natural history, being highly contagious and the aesthetic and psychotherapeutic effects of its treatment, the investigators intend to test the use of different concentrations of potassium hydroxide solution in the primary care setting.

METHODS:

A double blind, randomized clinical trial, in three groups of topic treatment is designed. The intended treatment consists on a daily application of potassium hydroxide in aqueous solution at 10% and 15% concentration, versus a placebo administered to the control group. 4 follow-up visits (15, 30, 45 and 60 days) are planned to evaluate treatment effectiveness and tolerance.

The main target of the trial is to determine the healing rate, defined as lesion disappearance in the affected zones after the topic application of the treatment. Secondary targets are the main characteristics and evolution of the affected zone (surface, number of lesions, size and density) description, tolerance evaluation (hyperpigmentation, itching, burning, pain), recurrence rate estimation and natural evolution of lesions in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Who are diagnosed with a molluscum contagiosum (MC) infection (clinical diagnosis).
* Who are between the ages of two and six.
* Whose parents or guardians have provided written informed consent for participation.

Exclusion Criteria:

* Immunocompromised patient (congenital or acquired).
* Patient has received other topical treatment within the last month.
* Patient has lesions on face, neck or genital area.
* Patient who, in the view of the attending physician, will not comply with treatment and/or scheduled visits.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Efficacy (diseappearance of lesions) | 60 days

CONTACTS AND LOCATIONS:
Locations (1):
- CAP Rambla Ferran, Lleida, Catalonia, Spain

REFERENCES:
- [Derived] Marsal JR, Cruz I, Teixido C, Diez O, Martinez M, Galindo G, Real J, Schoenenberger JA, Pera H. Efficacy and tolerance of the topical application of potassium hydroxide (10% and 15%) in the treatment of molluscum contagiosum: randomized clinical trial: research protocol. BMC Infect Dis. 2011 Oct 19;11:278. doi: 10.1186/1471-2334-11-278. PMID 22011376